CLINICAL TRIAL: NCT02783703
Title: Evaluation of Medium Chain Triglycerides in a Mixed Racial Population of Patients: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Caroline Apovian, BMC Faculty, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-35267
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Insulin Resistance
Keywords: Hyperinsulinemia
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCT (Experimental): Medium chain triglyceride (MCT) oil ingested daily for 6 weeks
  Interventions: Dietary Supplement: Medium chain triglycerides (MCT)

INTERVENTIONS:
Dietary Supplement: Medium chain triglycerides (MCT) — Subjects will consume 30 grams per 2000 kilocalories daily of medium chain triglyceride oil by mouth

SUMMARY:
The study team will investigate the racial differences in the metabolic and clinical responses to Medium chain triglycerides (MCT) between African American and Caucasian American subjects.

DETAILED DESCRIPTION:
It is generally accepted that type 2 diabetes (T2D) arises from the progression of insulin resistance (IR), with hyperinsulinemia (HI) as a compensatory response. The possibility that HI can precede and contribute to insulin resistance (IR) and metabolic syndrome (MS) has been suggested but not tested in humans. While IR and HI are closely associated, demonstrating a primary role for HI in T2D is key to the development of new treatment strategies for this disease. One group in which HI could play a bigger role in T2D is African Americans (AA) who are known to be more hyperinsulinemic than Caucasian Americans (CA). Racial disparities in T2D treatment outcomes adversely affect AA. Our main hypothesis is that suppression of HI will contribute to the prevention and treatment of T2D, especially among AA. Our goal in this pilot study is to show that consumption of medium chain triglycerides (MCT) in the diet will decrease basal insulin secretion and HI, and will lead to improvement in the insulin sensitivity index (Si). 24 subjects (12 AA, 12 CA) will participate in a clinical trial in which they will receive MCT for 6 weeks. Insulin secretion dynamics and insulin sensitivity will be assessed by use of the frequently sampled intravenous glucose tolerance test (FSIVGTT) and Bergman's minimal model analysis.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Males and female ambulatory subjects
* Self-identify as Caucasian/White or Black/African American
* Body Mass Index <=45

Exclusion Criteria:

* Diagnosis of type 2 diabetes or hemoglobin A1c >6.5
* Use of insulin, oral hypoglycemic, agents, or insulin-sensitizing agents
* Daily use of oral steroids
* Unstable weight within 3 months prior to baseline (e.g., weight gain or loss of >3%)
* Use of any weight loss medications or sex hormone therapy
* Daily use of psychotropic medications (for schizophrenia, bipolar disorder, obsessive compulsive disorder, posttraumatic stress disorder, psychotic disorder, mania)
* Chronic kidney disease, on dialysis or history of renal transplant
* Poorly controlled cardiovascular disease or congestive heart failure
* Severe peripheral vascular disease or severe liver disease
* Cancer
* A condition requiring use of oxygen such as severe chronic obstructive pulmonary disease
* Women who are pregnant, lactating, or actively trying to become pregnant
* Any cognitive or other disorders that may interfere with participation or ability to follow restrictions
* Abnormal TSH levels (<0.01 or >1.5x the upper limit)
* Weight >450 lb (205 kg) or height > 6'6"
* Severe claustrophobia
* Has had or is preparing for bariatric surgery (pre- or post-bariatric)
* Medically required use of anticoagulant therapies
* Current use of MCT oil
* Anemia (hemoglobin and/or hematocrit outside sex-specific normal ranges)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity to 6 weeks as measured by intravenous glucose tolerance test | Baseline to 6 weeks

SECONDARY OUTCOMES:
Change from baseline to 6 weeks in resting energy expenditure (kilocalories) | Baseline to 6 weeks
Change from baseline to 6 weeks in body composition (% fat, muscle and bone) | Baseline to 6 weeks
Change baseline to 6 weeks in physical activity (minutes of moderate or vigorous activity performed) | Baseline to 6 weeks
Assessment of the following from Baseline to end of intervention: Adverse Events (AEs), Vital Signs, Anthropometrics | Baseline to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Apovian, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Patient data is protected by HIPAA. Results will be published in a peer-reviewed journal.